CLINICAL TRIAL: NCT06453122
Title: Effect of Toothbrushing Without Chlorhexidine on Oral Hygiene Indices and Risks of Systemic Complications in Patients With Orotracheal Intubation: Randomized Pilot Clinical Study and Cost-effectiveness Analysis.
Brief Title: Effect of Toothbrushing Without Chlorhexidine on Oral Hygiene Indices in Patients With Orotracheal Intubation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5736-23
Record Dates: First submitted 2024-06-07; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-03

CONDITIONS: Oral Hygiene; Intensive Care; Chlorhexidine
MeSH Terms: interventions — Dental Care Team

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine (Active Comparator): patients with oral hygiene performed with tooth brushing and washing with 0.12% chlorhexidine
  Interventions: Other: Oral care
- Water (Sham Comparator): patients with oral hygiene performed with tooth brushing and washing with filtered water.
  Interventions: Other: Oral care

INTERVENTIONS:
Other: Oral care — The intervention group procedure will be carried out in the same way and frequency of the control group, however, replacing the chlorhexidine solution 0.12% for mineral water. Oral hygiene will be carried out by the nursing team, which will be blind to the indices to be evaluated. The team will be previously trained to carry out hygiene procedures by the team of ICU dental surgeons.

SUMMARY:
The oral hygiene method commonly used in intubated patients orotracheal is tooth brushing (mechanical removal) and washing the oral cavity and the orotracheal tube (TOT) with digluconate solution chlorhexidine (CLX). However, recent studies have demonstrated that the use of CLX in these conditions may expose the patient to a potential increased risk of mortality. Recent recommendations made by international bodies related to hospital biosafety no longer include the use of CLX in ICU oral hygiene routine. A question not yet answered in the literature is whether the absence of CLX in the critical patient's oral hygiene routine predisposes increased accumulation of dental plaque or microbial colonization related to the risk of systemic complications, such as pneumonia and sepsis. The cost-effectiveness of this protocol change also needs to be evaluated, as the withdrawal of CLX may result in changes in the risk profile morbidity and mortality during hospitalization. The present study aims to investigate whether brushing the oral cavity with mineral water changes the pattern of biofilm accumulation and clinical appearance of the oral mucosa in relation to brushing done with CLX. Microbiological analysis of the oropharyngeal biofilm and cost-effectiveness impact assessment will also be carried out.

DETAILED DESCRIPTION:
* Chlorhexidine group: Oral hygiene will be carried out in accordance with the standard operating procedures already carried out for all patients admitted to the ICU. First, the secretion contained in the oral cavity will be aspirated with a suction probe or a dental sucker or the suction brush itself before starting the oral hygiene procedure. The hygiene process will begin by moistening the oral cavity, using non-sterile gauze soaked in filtered mineral water and applying it to the entire oral mucosa. Subsequently, the sucking toothbrush or oral swab should be moistened frequently with 0.12% chlorhexidine digluconate solution and proceed with cleaning the dental surfaces on their buccal, palatal and occlusal surfaces, moving towards the oral cavity and tongue, using the bristle part of the toothbrush; With the region opposite the dental bristles or oral swab, the 0.12% chlorhexidine solution will be applied to the oral mucosa, palate, tongue dorsum and orotracheal tube, always performing a postero-anterior movement and removing any dirt with the aid of moistened gauze . The oral cavity will be constantly vacuumed throughout the oral hygiene procedure. Finally, the lips will be lubricated with a standardized lip moisturizer. The procedure will be carried out every 8 hours, that is, three times a day.
* Water group: The intervention group procedure will be carried out in the same way and frequency as the control group, however, replacing the 0.12% chlorhexidine solution with mineral water. Oral hygiene will be carried out by the nursing team, who will be blind to the indices to be evaluated. The team will be previously trained to carry out hygiene procedures by the ICU team of dental surgeons.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the adult ICU;
* age over 18;
* both sexes;
* orotracheal intubation monitored from the first day;
* absence of foci of infection in the oral cavity (periapical lesions,
* periodontal abscesses, extensive cavities, opportunistic infections);
* presence of at least five teeth per dental arch

Exclusion Criteria:

* patients in whom oral hygiene is not possible;
* patients extubated before 24 hours from baseline;
* patients with foci of infection in the oral cavity present in the baseline moment;
* patients who died before 24 hours from baseline;
* patients whose guardians do not authorize the research to be carried out;
* patients whose information about oral and general health and other study variables are not available in the medical record, are doubtful or not capable of collection.
* patients after heart surgery
* patients with reintubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Analyze oral cavity brushing | T0 (baseline) - first day of intubation; • T1 - after 3 days of intubation or immediately after extubation (with a minimum of 1 day of intubation); • T2 - after 7 days of intubation (if you still remain intubated).
  Analyze oral cavity brushing done with mineral water in the ICU in regarding the accumulation of biofilm and the appearance of the oral mucosa and compare these variables with brushing done with CLX.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda de P Eduardo, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klompas M, Branson R, Cawcutt K, Crist M, Eichenwald EC, Greene LR, Lee G, Maragakis LL, Powell K, Priebe GP, Speck K, Yokoe DS, Berenholtz SM. Strategies to prevent ventilator-associated pneumonia, ventilator-associated events, and nonventilator hospital-acquired pneumonia in acute-care hospitals: 2022 Update. Infect Control Hosp Epidemiol. 2022 Jun;43(6):687-713. doi: 10.1017/ice.2022.88. Epub 2022 May 20. PMID 35589091
- [Background] Klompas M, Branson R, Eichenwald EC, Greene LR, Howell MD, Lee G, Magill SS, Maragakis LL, Priebe GP, Speck K, Yokoe DS, Berenholtz SM. Strategies to prevent ventilator-associated pneumonia in acute care hospitals: 2014 update. Infect Control Hosp Epidemiol. 2014 Sep;35 Suppl 2:S133-54. doi: 10.1017/s0899823x00193894. No abstract available. PMID 25376073
- [Background] Prendergast V, Kleiman C, King M. The Bedside Oral Exam and the Barrow Oral Care Protocol: translating evidence-based oral care into practice. Intensive Crit Care Nurs. 2013 Oct;29(5):282-90. doi: 10.1016/j.iccn.2013.04.001. Epub 2013 May 20. PMID 23702324
- [Background] Bellissimo-Rodrigues WT, Menegueti MG, de Macedo LD, Basile-Filho A, Martinez R, Bellissimo-Rodrigues F. Oral mucositis as a pathway for fatal outcome among critically ill patients exposed to chlorhexidine: post hoc analysis of a randomized clinical trial. Crit Care. 2019 Nov 27;23(1):382. doi: 10.1186/s13054-019-2664-6. No abstract available. PMID 31775844
- [Background] Zhao T, Wu X, Zhang Q, Li C, Worthington HV, Hua F. Oral hygiene care for critically ill patients to prevent ventilator-associated pneumonia. Cochrane Database Syst Rev. 2020 Dec 24;12(12):CD008367. doi: 10.1002/14651858.CD008367.pub4. PMID 33368159